CLINICAL TRIAL: NCT06376773
Title: Neoadjuvant Treatment Based on Gastric Cancer Molecular Subtyping: Chemotherapy, Immunotherapy, or Targeted Therapy? -A Retrospective Real-World Data Analysis
Brief Title: Neoadjuvant Treatment Based on Gastric Cancer Molecular Subtyping.
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Fujian Medical University, Fujian Medical University
Other Study IDs: 2022KY123
Record Dates: First submitted 2024-04-15; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Gastric Cancer; Neoadjuvant Therapy; Multi-omics Analysis
MeSH Terms: interventions — Drug Therapy, Combination; apatinib; camrelizumab; Metabolic Networks and Pathways; Congresses as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- mesenchymal: Based on RNA-seq transcriptome, patients were divided into mesenchymal, and received neoadjuvant chemotherapy with apatinib or not
  Interventions: Procedure: combination chemotherapy with Apatinib or Camrelizumab
- immunogenic: Based on RNA-seq transcriptome, patients were divided into immunogenic, and received neoadjuvant chemotherapy with Camrelizumab or not
  Interventions: Procedure: combination chemotherapy with Apatinib or Camrelizumab
- metabolic: Based on RNA-seq transcriptome, patients were divided into metabolic, and received neoadjuvant chemotherapy with apatinib, Camrelizumab or not
- classic: Based on RNA-seq transcriptome, patients were divided into classic, and received neoadjuvant chemotherapy with apatinib, Camrelizumab or not

INTERVENTIONS:
Procedure: combination chemotherapy with Apatinib or Camrelizumab — Apatinib, chemotherapy alone, Camrelizumab
  Other Names: mesenchymal; immunogenic; metabolic; classic
  Groups: immunogenic; mesenchymal

SUMMARY:
Extensive research employing diverse omics methodologies has unveiled a varied landscape of gastric cancer (GC). Recent progress in next-generation sequencing and other genomic technologies has facilitated a more intricate exploration of GC at the molecular level. This study aimed to identify the most effective drug therapeutics for patients with the mesenchymal subtype of gastric cancer.Based on RNA-seq transcriptome, 234 patients were divided into four molecular subtypes: mesenchymal, immunogenic, metabolic, and classic.Our analysis has revealed that, for neoadjuvant therapy in advanced gastric cancer (AGC), the mesenchymal subtype stands out as the ideal patient population benefiting from Apatinib, without a concurrent increase in postoperative complications.

DETAILED DESCRIPTION:
The advent of immunotherapy and targeted therapies has recently provided new options for AGC treatment. However, not all patients benefit from immunotherapy or targeted therapy, resulting in unsatisfactory overall treatment outcomes during the perioperative period. An ineffective treatment imposes significant financial burden, causes drug-related side effects that deteriorate their quality of life, and potentially delays subsequent treatment.

Evaluate the objective response rate (ORR) of the combination of camrelizumb, apatinib, and neoadjuvant chemotherapy for the treatment of advanced gastric patient Median survival time (OS);

Disease free survival time (DFS);

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with gastric adenocarcinoma and received neoadjuvant therapy

Exclusion Criteria:

* Patients with distant metastases, gastric stump cancer, or missing neoadjuvant chemotherapy data were excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study collected data from 234 patients diagnosed with gastric adenocarcinoma at Fujian Medical University Union Hospital (FMUUH) who underwent gastrectomy after receiving neoadjuvant therapy (NAT) between January 2019 and January 2022.
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
overall survival | 2years
  overall survival

SECONDARY OUTCOMES:
objective response rate | 6months
  objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fuji'an, China

IPD SHARING:
Plan to Share IPD: No